CLINICAL TRIAL: NCT05017155
Title: A Phase III, Randomised, Double Blinded, Head-to-head, Single-site, Cross-over Trial of Lamotrigine Versus Mexiletine for Non-dystrophic Myotonias
Brief Title: MExiletine Versus Lamotrigine in Non-Dystrophic Myotonias
Acronym: MEND
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18/0582
Record Dates: First submitted 2021-08-11; First posted 2021-08-23 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Non-Dystrophic Myotonia
MeSH Terms: interventions — Mexiletine; Lamotrigine; Tablets

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from University College London Hospital (UCLH). After screening and consent, randomisation will occur to one of two arms. The participant will participate in two consecutive time periods. A time period will consist of 8 weeks of Mexiletine or Lamotrigine. The second time period will then occur after 7 days of washout. The patient will then take the alternative drug. Visits will occur at the end of each period and can be undertaken remotely as required. At each visit, the Interactive Voice Response (IVR)-Diary score will be performed and secondary measures including the Brief Pain Inventory, Modified Fatigue Severity Scale and Medical Outcomes Study Questionnaire (SF-36). Objective recordings including Timed up and Go (TUG), Timed Sit to Stand (TST). Safety data will be recorded simultaneously. A participant diary will be utilised to record daily IVR-Diary scores, medication compliance and activity measures.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lamotrigine (Active Comparator): When on the lamotrigine treatment arm, the participant will commence at lamotrigine 25mg (milligram) daily for two weeks; then increase to 25mg twice daily for two weeks; then increase to 50mg daily for one week; then increase to 100mg in the morning, 50mg at midday and 50mg at night for one week; then increase to 100mg in the morning, 50mg at midday and 100mg at night for two weeks.
  Interventions: Drug: Mexiletine; Drug: Lamotrigine 25Mg Oral Tablet, Extended Release
- Mexiletine (Active Comparator): When on the mexiletine treatment arm, the participant will commence at mexiletine 100mg daily for two weeks; then increase to 200mg daily for two weeks; then increase to 200mg twice daily for one week; then increase to 200mg three times a day for one week; then remain on 200mg three times a day for two weeks.
  Interventions: Drug: Mexiletine; Drug: Lamotrigine 25Mg Oral Tablet, Extended Release

INTERVENTIONS:
Drug: Mexiletine — Mexiletine is a sodium channel blocker shown to be effective in reducing myotonia in a multi-centre randomised trial.
Drug: Lamotrigine 25Mg Oral Tablet, Extended Release — Lamotrigine is an alternative sodium channel blocker that has been shown to be effective in one randomised controlled trial. It is currently used as a licensed medication for other neurological conditions.

SUMMARY:
This is a clinical trial to determine if Lamotrigine is non-inferior to Mexiletine for the treatment of myotonia in patients with Non-Dystrophic Myotonia.

Non-dystrophic Myotonia is a genetic condition for which there is no cure. It affects patients for the duration of their life and impacts work, leisure and can lead to significant morbidity.

The study is a cross-over design - participants will be randomized to either lamotrigine or mexiletine first for 8 weeks and then swap over after a week wash-out to the other medication for a further 8 weeks. Participants and investigators will be blinded to the treatment schedule. 60 participants will recruited through the clinical service, national registry and national liaison.

DETAILED DESCRIPTION:
The current first line treatment for Non-Dystrophic Myotonia (NDM) - Mexiletine - is ineffective in some patients, cannot be used in pregnancy, has side effects and is expensive with limited access in the UK, prompting the clear need for an alternative. A recent open label trial has demonstrated efficacy of Lamotrigine in treating NDMs, raising the possibility of Lamotrigine superseding Mexiletine as the first line agent. As the nationally commissioned highly specialised service for channelopathies, more patients are being seen than in other centres, have a track record of trials in NDMs published in high impact factor journals, and are best placed to conduct a trial of Mexiletine versus Lamotrigine.

Clinical morbidity: NDM impairs mobility, causes social embarrassment and impacts on quality of life. NDMs are a group of rare genetic neuromuscular disorders caused by dysfunction of ion channels that are critical for muscle membrane excitability. The hallmark of these disorders is that symptoms occur in an episodic or paroxysmal fashion causing acute disability. The NDMs include myotonia congenita (MC), sodium channel myotonia (SMC) and paramyotonia congenita (PMC). They have a point prevalence in England of 1.12/100,000. MC is due to mutations in the Chloride Channel gene (CLCN1), which codes for the muscle chloride channel clc-1. SMC and PMC are caused by mutations in the Sodium Channel Gene (SCN4A), which codes for the skeletal muscle voltage gated sodium channel Nav1.4. Both of these channels are essential for regulating normal muscle membrane excitability, muscle contraction and relaxation. NDMs are therefore unified by a common pathomechanism of altered muscle membrane excitability. The membrane becomes hyper-excitable resulting in spontaneous depolarisation and contraction after a motor nerve stimulus.

The primary clinical manifestation of NDM is myotonia - delayed relaxation of skeletal muscle after contraction. Myotonia is experienced by patients as muscles "locking", "sticking" or "cramping". Symptoms commonly affect the leg muscles and are precipitated by sudden or initial movement leading to falls and injury. They are also exacerbated by prolonged sitting, especially after preceding physical activity, and changes in environmental temperature. This can be particularly problematic on public transport which may stop abruptly, causing falls or inability to exit quickly enough, missing their destination. These difficulties can limit independence, social activity, choice of employment and are often socially embarrassing. The symptomatic relationship with activity often leads to sedentary behaviour which in turn is a risk factor for additional co-morbidities e.g. heart disease or stroke. The condition is frequently painful, with pain and impaired physical ability impacting significantly on quality of life. Symptoms commonly worsen during pregnancy which can be compounded by the need to discontinue current pharmacological therapies due to a lack of safety data during pregnancy.

Limitations of current pharmacological therapies: There is currently no cure or disease-modifying treatment for NDM. Sodium channel blockers are used for symptomatic relief. Previously it was shown that Mexiletine is effective in reducing myotonia and improving quality of life in an international randomised placebo controlled trial. Mexiletine has become first line treatment for NDM but not all patients respond to mexiletine and a significant proportion, up to a third develop side effects, the most common being gastro-intestinal. Mexiletine has also been shown to be less beneficial for patients with MC than those with Sodium Channel Myotonia (SCM) or PMC. Additionally, mexiletine cannot be prescribed in pregnancy, when myotonia often worsens. Mexiletine is expensive and can only be accessed by specialist centres. This can have practical difficulties and limit access to treatment for some patients. There is a clear clinical need for an alternative therapeutic option to Mexiletine for the treatment of NDM.

The study design has been chosen specifically to allow participants to be internal controls. The degree of myotonia varies with changes in temperature and degree of activity. A highly active participant cannot be directly compared to a sedentary participant, hence the use of internal controls in an 'n of one' trial accounts for this variability.

The participants and investigators will be blinded with the use of over-encapsulated mexiletine and lamotrigine dispensed via a predetermined randomisation scheduled. Blinding is important to eliminate bias and in ensuring unbiased completion of subjective questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥ 18years),
* genetically confirmed non-dystrophic myotonia (NDM),
* presence of symptomatic myotonia as reported by the participant.

Exclusion Criteria:

* concomitant medical conditions that would preclude the use of mexiletine or lamotrigine,
* evidence of severe kidney disease or severe liver impairment [estimated glomerular filtration rate (eGFR) as calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Equation <60ml/min/1.73m2],
* pregnant or breastfeeding women,
* participation in other treatment studies <30days before enrolment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-04-02 (Estimated)

PRIMARY OUTCOMES:
Interactive Voice Response (IVR) -diary score | Time Frame: last two weeks of each treatment period - [Minimum value 0- no myotonia. Maximum value 9 - severe myotonia].
  Improvement seen on the 9 point Interactive Voice Response (IVR) -diary score

SECONDARY OUTCOMES:
Secondary Outcome - Timed up and go | end of each treatment period (two months)
  Timed up and go
Secondary Outcome - Timed sit to stand | end of each treatment period (two months)
  Timed sit to stand
Fatigue Scale | end of each treatment period (two months)
  minimum 9 - minimal fatigue. maximum 63 - severe fatigue
Secondary Outcome | end of each treatment period (two months)
  Brain Pain inventory
Short-Form Health Survey (SF-36) | end of each treatment period (two months)
  minimum score 0 - more disability; maximum score 100 - less disability
Myotonia Behaviour Score | end of each treatment period (two months)
  minimum score 0 - minimum stiffness; maximum score 5 - incapacitating stiffness

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Request for sharing anonymised data can be made to the Chief Investigator (CI) for discussion/consideration.

REFERENCES:
- [Derived] Vivekanandam V, Skorupinska I, Jayaseelan DL, Matthews E, Barohn RJ, McDermott MP, Hanna MG. Mexiletine versus lamotrigine in non-dystrophic myotonias: a randomised, double-blind, head-to-head, crossover, non-inferiority, phase 3 trial. Lancet Neurol. 2024 Oct;23(10):1004-1012. doi: 10.1016/S1474-4422(24)00320-X. PMID 39304240